CLINICAL TRIAL: NCT02026440
Title: Collection and Testing of Human Oral Fluid Samples/VioOne OF Sample Collection Device
Brief Title: Evaluation of An Oral Fluid Collection Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Avioq, Inc. (Industry)
Collaborators: Clinical Reference Laboratory, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 200008; FDA Pre-Submission Q130748 (Other: Avioq,Inc.)
Record Dates: First submitted 2013-12-12; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Smoking
Keywords: oral fluid collection device cotinine detection
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Smokers: Those who smoke at least one cigarette a day.
- Non smokers: Those who have not smoked for at least one week when the sample is collected.

SUMMARY:
The VioOne Oral Fluid Sample Collection Device can be used to collect human oral fluid samples for detection of cotinine using an ELISA cotinine assay.

DETAILED DESCRIPTION:
The Study to evaluate the VioOne Oral Fluid Sample Collection Device (herein referred to as VioOne Device) will consist of several sub-studies as described below:

A. Recovery Study

This study will determine the percent recovery of cotinine spiked into the oral fluid of non-smokers collected with the VioOne Sample Collection Device.

1. Sample collection

   Oral fluid will be collected per the VioOne package insert from five individuals self-reported to be non-smokers. The samples collected will then be individually spiked with cotinine to concentrations of 0, 5, 10, 15 or 25ng/mL. Two sets of each concentration will be prepared. One set will be stored at 2-8°C prior to testing and one set will be shipped per routine shipping conditions and tested upon return.
2. Testing

   Each sample will then be tested in duplicate with the Calbiotech Cotinine ELISA assay and the percent recovery will be calculated for each level by comparing the detected concentrations to the spiked concentrations.
3. Data Analysis Percent recovery will be calculated for each level by comparing the detected concentrations to the spiked concentrations.

B. Sensitivity/Accuracy Study The study goal is to show that the Calbiotech Cotinine ELISA is capable of distinguishing smokers from nonsmokers when oral fluid samples collected with the VioOne Sample Collection Device are used.

1. Sample Collection A minimum of two study sites will participate in this study. Approximately 218 individuals will be enrolled in this study. At least 58 collected samples must be from self-declared smokers. Oral fluid samples will be collected from individuals, who will give the informed consent and self-report in an anonymous fashion whether or not the individual is a smoker and number of cigarettes smoked per day on average. Two samples will be collected from each individual for this study. One sample will be collected using the VioOne Collection Device and one will be collected using a commercially available saliva collection cup.

   There will be no age, gender or race criteria for enrolling the patients.
2. Testing All samples collected with the VioOne Sample Collection Device will be tested with the Calbiotech Cotinine ELISA and the neat saliva samples collected with the saliva collection cups will be tested by GC/MS, the latter being the gold standard method.
3. Data Analysis The GC/MS results will be used as the gold standard for assessing the clinical sensitivity and specificity of the assay using oral fluid samples collected with the VioOne Oral Fluid Collection Device.

C. Assay Specificity Study Beverages and Household materials will be tested for interference in the detection of cotinine in oral fluid.

1. Sample Collection Oral Fluid samples will be collected from individuals self-reported as non-smokers and the resulting sample/buffer matrix will be pooled.

   The pool will be divided into 15 aliquots and individually spiked each of the following 14 compounds. One aliquot form the pool will remain un-spiked. Each spiked aliquot will then be further divided into three aliquots. One aliquot will remain spiked with the compound only, one aliquot will be further spiked with 5ng/mL of Cotinine and one aliquot will be further spiked with 15ng/mL Cotinine.
2. Testing Each sample will then be tested in duplicate.

   The following compounds will each be spiked at a final concentration of 10% unless otherwise noted:

   Sugar Water Alcohol (Ethanol) Toothpaste Whole Blood (10mg/mL) Cranberry Juice Hydrogen Peroxide Baking Soda Sodium Chloride Orange Juice Cola Cough Syrup Antiseptic Water Hemoglobin (10mg/mL)
3. Data Analysis Results will be compared to the expected performance as measured in the precision study. (the precision study does not require the use of collected human oral fluid)

D. Assay Specificity Study

The effect of potential food and other oral cavity contaminants will be evaluated in a timed study.

1. Sample Collection

   Ten individuals self-reported to be non-smokers will be recruited for this study.

   One sample will be collected using the VioOne Sample Collection Device from each individual immediately prior to the start of the study. Each individual will then be given a piece of hard candy to consume. Additional samples will be collected with VioOne immediately post consumption, ten minutes post consumption then every thirty minutes up to three hours.

   After all samples are collected each sample will be divided into two aliquots. One aliquot will be spiked with 5ng/mL cotinine and one aliquot will be spiked with 15ng/mL cotinine.
2. Testing Each sample/spike/time point will be tested in triplicate
3. Data Analysis Results will be compared to the expected performance as measured in the precision study. (the precision study does not require the use of collected human oral fluid)

E. Stability of sample in sample collection buffer A study will be performed to establish the stability of samples stored in sample collection buffer at various temperatures over time.

1. Sample Collection

   Oral Fluid samples will be collected from individuals self-reported as non-smokers and the resulting sample/buffer matrix will be pooled.

   The pool will be split into three aliquots. One aliquot will be spiked with 7.5ng/mL cotinine, one aliquot will be spiked with 10ng/mL cotinine and one aliquot will remain non-spiked.

   Each one of the spikes and the non-spike will be aliquoted into four tubes and stored at -20 oC, 2-8oC, room temperature and 37oC.
2. Testing

   Each sample will be tested in eight replicates at Day 0, 7, 14, 21, 28 and 35.
3. Data analysis

The sample is considered stable at the test time point when the 95% confidence interval for the cotinine concentration at a given day for the sample overlaps that of Day 0.

F. ELISA and Device Stability

A long term stability study will be performed to establish the stability and expiration dating of the Calbiotech Cotinine ELISA assay along with the VioOne Sample collection Device.

1. Sample Collection

   At each testing time point, samples from three individuals will be collected. Each individual will provide three samples- one with each of three lots of VioOne Sample Collection Devices.

   The resulting sample/buffer matrix obtained from each lot of VioOne Sample Collection Device will be pooled (a total of 3 individual samples per pool and a total of 3 pools).

   The resulting pools will then be divided into two aliquots. One aliquot will be spiked with 5ng/mL cotinine and 25ng/mL cotinine.
2. Testing

   Each spiked sample will be tested in eight replicates over a period of 21 months. Over the course of testing, three ELISA assay lots will be used.
3. Data Analysis

The Calbiotech Cotinine ELISA assay and the VioOne Sample Collection Device are considered stable when the samples tested at each time point produce results within the 95% confidence interval for the cotinine concentration overlaps that of Day 0.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults (aged 18 or older)

Exclusion Criteria:

* individuals with significant health problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and adult population
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Presence of Nicotine in Collected Oral Fluid Samples | Within one week of sample collection
  ELISA assay in comparison with the Mass-spec method will be used to detect the presence of nicotine in the oral fluid samples collected with the VioOne collection device.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Reddington, B.S., Study Chair — Avioq, Inc.
Locations (1):
- Avioq, Research Triangle Park, North Carolina, United States